CLINICAL TRIAL: NCT02576236
Title: Comparison of the Efficacy and Tolerance of Triple Therapy Guided by the PCR Detection of Clarithromycin Resistance WITH Empiric Concomitant Quadruple Therapy for Helicobacter Pylori Infection: a Randomised Multicentre Trial
Brief Title: Therapeutic Trial Comparing Triple Therapy Guided by the PCR Detection of Clarithromycin Resistance vs Empiric Concomitant Quadruple Therapy for Helicobacter Pylori Infection
Acronym: Hepysé
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140928; 2015-A00457-42 (Other: IDRCB)
Record Dates: First submitted 2015-09-30; First posted 2015-10-15 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: H Pylori Infection Eradication; Antibiotics Therapeutic Strategies; H Pylori Eradication
Keywords: Naïve patient; Suspicion of H pylori infection; Endoscopy; Antibiotics therapeutic strategies; Urea breath test
MeSH Terms: interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple therapy guided by result of the molecular resistance (Experimental): * If clarithromycin S : high dose PPI (Esoméprazole 40mg X 2/ d) - amoxicillin 1gX2 / d - clarithromycin 500mgX2 / d The total duration of treatment is 14 days.
  * If clarithromycin R: high dose PPI (Esoméprazole 40mg X 2/ d) - amoxicillin 1gX2 / d- levofloxacin 500mg X2 / d The total duration of treatment is 14 days.
  Interventions: Other: Triple therapy guided by the result of the molecular resistance test
- Quadruple concomitant therapy (Active Comparator): high dose PPI (Esoméprazole 40 mg X 2 / d- amoxicillin 1gX2 / d - - clarithromycin 500mgX2 / d - metronidazole 500mgX2 / d for 14 days
  Interventions: Other: Quadruple concomitant therapy treatment

INTERVENTIONS:
Other: Quadruple concomitant therapy treatment — Quadruple concomitant therapy treatment:
  high dose PPI (Esoméprazole 40 mg X 2 / d- amoxicillin 1gX2 / d - - clarithromycin 500mgX2 / d - metronidazole 500mgX2 / d for 14 days
  Other Names: therapeutic procedure
  Arms: Quadruple concomitant therapy
Other: Triple therapy guided by the result of the molecular resistance test — Triple therapy guided by the result of the molecular resistance test:
  * If clarithromycin S : high dose PPI (Esoméprazole 40mg X 2/ d) - amoxicillin 1gX2 / d - clarithromycin 500mgX2 / d The total duration of treatment is 14 days.
  * If clarithromycin R: high dose PPI (Esoméprazole 40mg X 2/ d) - amoxicillin 1gX2 / d- levofloxacin 500mg X2 / d The total duration of treatment is 14 days.
  Other Names: therapeutic procedure
  Arms: Triple therapy guided by result of the molecular resistance

SUMMARY:
The H pylori infection remains a public health problem. The eradication rate with the first line triple therapy (PPI-amoxicillin-clarithromycin) is insufficient (estimated at 70%) due to the frequency of resistance to clarithromycin, which reaches 21% in France. Until now,European and French consensus recomended tofavor sequential therapy (5 days PPI-amoxicillin and 5 days PPI-clarithromycin-metronidazole) or quadruple bismuth therapy ( 10 days PPI-tetracyclin,-metronidazole- bismuth). Studies in countries with low prevalence of clarithromycin resistance reported eradication rate of 85% with sequential therapy and reported a low impact of clarithromycin resistance on the effectiveness of this treatment. However, recent studies suggest a greater impact of clarithromycin resistance. Recent meta-analysis shows that empiric sequential therapy is less efficacious than concomitant quadruple therapy. Therefore, recent Maastricht V / Florence meeting October 7-8 2015) recommended to abandon sequential therapy and to favor 14 days concomitant therapy in first line in order to reach an eradication rate >90%.

In a multicenter randomized clinical trial (HELICOSTIC 2010-2011 AO ICST 2009), we compared a triple therapy guided by the results of a PCR test that detects resistance to clarithromycin and levofloxacin (HelicoDR ®) to empirical triple therapy (PPI-amoxicillin-clarithromycin). 1384 patients and among them 526 infected patients were enrolled in 10 centers. The results in 415 patients were 73.1% for the empirical treatment versus 85.5% (p <0.001) for the treatment guided by PCR HelicoDR®. This study also demonstrated the limits of the test HelicoDR®: onerous, possibility of contamination, little practical contribution of the determination of resistance to quinolones.

Moreover, it has been shown that triple therapy efficiency could be optimized by increasing duration up to 14 days and increasing dose of PPI to 40mg b.d;.and eradications rates > 90% were reported with susceptible to clarithromycin strains.

Adverse events are less common with optimized triple therapy than with concomitant quadruple therapy.

The main objective is to compare the efficacy of optimized triple therapy guided by the results of a PCR test (eradication rates 90% hypothesized) with quadruple concomitant therapy (eradication rate 90% hypothesized).

The secondary objective is to determine side effects of optimized guided triple therapy as well as the quadruple concomitant therapy in France.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Hospitalized or out-patients referred to one of the participating centers for upper gastrointestinal endoscopy
* Who did not received a previous eradication treatment
* Willing to participate and signed inform consent. Finally only patients with bacteriologically documented H. pylori infection (PCR) will be included.

Exclusion Criteria:

* Patient having already been treated to eradicate H pylori
* No affiliation to social insurance
* Person under legal protection
* Refusal for signing informed consent
* Patient included in another trial with medication
* Patient unable to take oral medication ongoing
* Patient with severe life-threatening disease in the short term
* Contraindication to the PPIs, amoxicillin, metronidazole, clarithromycin, levofloxacin, tetracyclin or bismuth
* Patient under treatment with antibiotics or PPI without possibility of interruption for 4 weeks
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Eradication rate on the basis of a negative C13 - urea breath test done 6-12 weeks after the end of treatment | at 34 month
  Eradication rates will be compared between the patients allocated to standard treatment currently recommended (quadruple concomitant treatment, control group) and patients allocated to triple therapy chosen according to the results of molecular detection of clarithromycin resistance (guided triple therapy,, test group). The breath test is recognized as a sensitive and specific test for infection with H. pylori, particularly in the context of monitoring the efficacy of treatment. It will be carried out blindly to allocated group.

SECONDARY OUTCOMES:
Safety criteria will include all adverse events occurring in the two treatment groups | at 34 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Delchier, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Amiot A, Hacoon J, Heluwaert F, Mion F, Lamarque D, Moussata D, Mimouni M, Delchier JC, Durand-Zaleski I, Audureau E, Bastuji-Garin S; HEPYSE Study Group. 14-day tailored PCR-guided triple therapy versus 14-day non-Bismuth concomitant quadruple therapy for Helicobacter pylori eradication: A multicenter, open-label randomized noninferiority controlled trial. Helicobacter. 2024 Mar-Apr;29(2):e13076. doi: 10.1111/hel.13076. PMID 38680067